CLINICAL TRIAL: NCT00244049
Title: "Primary Care Alcohol Intervention in College Students"
Brief Title: CHIPs or College Health Intervention Projects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 1R01AA014685-01 (NIH); 1R01AA014685-01 (NIH)
Record Dates: First submitted 2005-10-21; First posted 2005-10-25 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Counseling; Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brief clinician advice (Experimental)
  Interventions: Behavioral: counseling; Other: Brief Intervention

INTERVENTIONS:
Behavioral: counseling — Physicians discussed high-risk/binge drinking with college-aged individuals in a health care setting.
Other: Brief Intervention — Physicians discussed effects of high-risk/binge drinking with college-aged individuals in a health care setting.

SUMMARY:
The goal of the study is to test the efficacy of brief clinician advice in reducing the frequency of high-risk drinking and alcohol-related harm in a population of college students seeking care at five university health care clinics. High-risk drinking is defined as 1) 8 or more episodes of heavy drinking (5 or more drinks in a row) in the past 28 days for male and female students, and/or 2) 50 drinks for male and 40 drinks for female students in the past 28 days, and/or 3) 15 drinks for male and 12 drinks for female students in the past 7 days, and/or 4) One or more episode(s) of heavy drinking which includes 15 or more drinks in a row.

ELIGIBILITY:
Inclusion Criteria:

* subjects who screen positive for high risk drinking on the Health Screening Survey (HSS) and Baseline interview

Exclusion Criteria:

* Students who will be leaving campus due to graduation or for an extended absence prior to the first face to face intervention Female students who are pregnant at the time of randomization Students who are currently suicidal at the time of the baseline interview Students under 18 years of age Students who drink more than 200 drinks in 28 days (referred for treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2004-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Reduction in binge/high-risk drinking in college-aged students. | 6-months

SECONDARY OUTCOMES:
c) fr. of accidents, d) fr. of campus vandalism and interaction police; e) academic perf; f) fr. of unwanted sex; g) fr. of high-risk sex; h) fr. of physical altercations i) ER visits and hospital days; and j) cost vs. benefit of the intervention. | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fleming, MD, Principal Investigator — University of Wisconsin, Madison